CLINICAL TRIAL: NCT02131519
Title: Utility of Ultrasonography During Internal Jugular Vein Catheterisation in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, specialist anesthesiologist, Ankara University
Other Study IDs: 13968; USG13968
Record Dates: First submitted 2014-05-04; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Number of Trials; Complication Rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- internal jugular vein catheter: pediatric patients required internal jugular vein catheter
  Interventions: Procedure: internal jugular vein catheter placement

INTERVENTIONS:
Procedure: internal jugular vein catheter placement

SUMMARY:
Central venous access may be essential in pediatric patients for fluid and a blood product administration, medication, parenteral nutrition, renal replacement therapy and hemodynamic monitoring. Obtaining central venous access in pediatric patients can be challenging, failure rates in pediatric patients range from 5% to 19% with reported complication rates from 2,5% to 22% The landmark technique has been standard approach for many years. In comparison with landmark method in pediatric patients the use of ultrasound is associated with an increased success rate decreased operative time, reduced number of cannulation attempts , and a decreased number of carotid artery punctures. We wanted to evaluate our success rate using ultrasound as a guidance during central vein insertion.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients required internal jugular vein catheter

Exclusion Criteria:

* aged smaller than 1 month

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients aged more than 1 month
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
success rate | during anesthesia

SECONDARY OUTCOMES:
complication rate | during anesthesia

OTHER OUTCOMES:
effect of experience | during anesthesia

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University, Pediatric Surgery, Ankara
  - Ankara University, Ankara